CLINICAL TRIAL: NCT07084337
Title: Effects of a Bodypump Training Program on Resting Blood Pressure and Physical Fitness in Sedentary Older Adults With Hypertension
Acronym: BPFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Manuel Jesús Rodríguez Chavarría, PhD Student, Universidad de Extremadura
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP-AH-FIT
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Older Adults; Functional Capacity; Resistance Training
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bodypump Group (Experimental)
  Interventions: Behavioral: Bodypump Training Program
- Group Control (No Intervention)

INTERVENTIONS:
Behavioral: Bodypump Training Program — Participants in this group performed a structured 8-week Bodypump program consisting of three sessions per week (Monday, Wednesday, and Friday), each lasting 45 minutes. The sessions followed the official Les Mills format, incorporating choreographed resistance exercises using barbells, weight plates, and a step platform. All movements were synchronized with music and led by certified instructors. Participants completed high-repetition, low-load exercises (~20% of 1RM) targeting major muscle groups. Exercises were adapted to individual capabilities to ensure safety and promote adherence.
  Arms: Bodypump Group

SUMMARY:
This study aimed to evaluate the effects of an eight-week Bodypump® group training program on resting blood pressure and physical fitness in sedentary older adults with hypertension. Bodypump is a choreographed resistance exercise class performed in groups, guided by certified instructors, and accompanied by music. It uses light weights and high repetitions, making it accessible and engaging for older individuals.

Thirty-two participants aged 55 and older with a medical diagnosis of hypertension were randomly assigned to either an intervention group (Bodypump classes, 3 times per week for 8 weeks) or a control group that maintained their usual sedentary behavior.

The main outcome was resting blood pressure (systolic and diastolic). Secondary outcomes included measures of functional fitness assessed using the Senior Fitness Test (SFT) battery: lower and upper body strength, aerobic endurance, agility, and balance.

Results showed a significant reduction in systolic and diastolic blood pressure in the Bodypump group compared to the control group. Participants also experienced significant improvements in physical performance measures.

This study suggests that structured group-based resistance training programs such as Bodypump are an effective non-pharmacological intervention for improving cardiovascular health and functional fitness in older adults with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age over 55 years
* Clinical diagnosis of hypertension
* Sedentary lifestyle for the past six months
* Medical clearance to participate in supervised physical activity
* Minimum functional fitness to perform testing and Bodypump exercises

Exclusion Criteria:

* Orthopedic or cardiovascular conditions that contraindicate physical exercise
* Unstable or uncontrolled hypertension
* Participation in any other structured exercise programme during the intervention
* Inability to perform the functional tests or Bodypump sessions safely

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Resting Blood Pressure (Systolic and Diastolic) | Baseline and 8 weeks of intervention.
  Change in systolic and diastolic blood pressure measured using an Omron M3 Intellisense automatic monitor. Measurements were taken at baseline and at 8 weeks, following standardized procedures.
Resting Blood Pressure | Baseline and 8 weeks of intervention.
  Change in systolic and diastolic blood pressure measured using an Omron M3 Intellisense automatic monitor. Measurements were taken at baseline and at 8 weeks, following standardized procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Osuna fitness, Osuna, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided